CLINICAL TRIAL: NCT05581719
Title: A Phase 1/2a Study Evaluating Allocetra-OTS as Monotherapy or in Combination With Anti-PD-1 Therapy for the Treatment of Advanced Solid Tumor Malignancy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Enlivex Therapeutics RDO Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ENX-CL-04-002a
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor; Peritoneal Metastases; Peritoneal Cancer
MeSH Terms: interventions — Nivolumab; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage 1 (Allocetra-OTS monotherapy) (Experimental): Dose escalation of Allocetra-OTS up to 10 x 10^9 cells by IV or IP administration.
  Interventions: Drug: Allocetra-OTS
- Stage 2.1 (Allocetra-OTS in combination with anti-PD-1 therapy) (Experimental): Dose escalation of Allocetra-OTS up to 10 x 10^9 cells by IV or IP administration, with IV nivolumab 240 mg.
  Interventions: Drug: Allocetra-OTS; Drug: Nivolumab
- Stage 2.2 (Allocetra-OTS in combination with anti-PD-1 therapy) (Experimental): Dose escalation of Allocetra-OTS up to 10 x 10^9 cells by IV or IP administration, with IV tislelizumab 200 mg.
  Interventions: Drug: Allocetra-OTS; Drug: Tislelizumab

INTERVENTIONS:
Drug: Allocetra-OTS — Allocetra-OTS is a cell-based therapy consisting of non-HLA matched allogeneic peripheral blood mononuclear cells, derived from a healthy human donor following a leukapheresis procedure, induced to an apoptotic stable state.
Drug: Nivolumab — Immune checkpoint inhibitor (anti-PD-1 antibody)
  Arms: Stage 2.1 (Allocetra-OTS in combination with anti-PD-1 therapy)
Drug: Tislelizumab — Immune checkpoint inhibitor (anti-PD-1 antibody)
  Arms: Stage 2.2 (Allocetra-OTS in combination with anti-PD-1 therapy)

SUMMARY:
This is an open-label, non-randomized, multicenter, Phase 1/2a study to evaluate the safety and potential efficacy of Allocetra-OTS in the treatment of advanced solid tumor malignancy as monotherapy or in combination with an anti-PD-1 therapy.

DETAILED DESCRIPTION:
Despite the advent of novel targeted and immunotherapeutics for the treatment of solid tumors, many patients remain without cure.

Allocetra-OTS is an immunomodulatory cell-based therapy consisting of allogeneic peripheral blood mononuclear cells that have been modified to be engulfed by macrophages and reprogram them into their homeostatic state.

This is an open-label, non-randomized, multicenter, Phase 1/2a study to evaluate the safety and potential efficacy of Allocetra-OTS in the treatment of advanced solid tumor malignancy as monotherapy (Stage 1), and in combination with an anti-PD-1 therapy (Stage 2).

Allocetra-OTS will be administered systemically or locally (intravenous [IV] or intraperitoneal [IP]) according to the tumor location.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed locally advanced, unresectable or metastatic solid tumors, that have relapsed or have been refractory to available approved therapies, or patients who are not eligible for or declined additional standard of care systemic therapy.

   Patients with peritoneal carcinomatosis can be eligible if an appropriate IP catheter or port can be placed.
2. Patients must have measurable disease.
3. Age ≥ 18 years old.
4. ECOG performance status ≤1.
5. Adequate renal function, hepatic function, and bone marrow function.

Exclusion Criteria:

1. Primary central nervous system (CNS) malignancy or CNS involvement, unless stable clinically.
2. Clinically significant uncontrolled infection, autoimmune or inflammatory diseases requiring systemic immunosuppression, clinically significant cardiovascular disease, severe pulmonary diseases or additional malignancies.
3. [For patients in Stage 2] Patients who previously experienced an ICI-related adverse reaction that resulted in discontinuation of the ICI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Safety of Allocetra-OTS | 3-5 weeks
  Characterize the safety of Allocetra-OTS based on the dose-limiting toxicities (DLTs) of Allocetra-OTS as monotherapy or in combination with anti-PD1 therapy.

SECONDARY OUTCOMES:
Overall Response Rate (ORR)/Best Overall Response Rate (BORR) | 12 months
  Overall Response Rate (ORR)/Best Overall Response Rate (BORR) (percentage of patients who achieve best response of complete response [CR] or partial response [PR]).
Clinical benefit rate (CBR) | 12 months
  Clinical benefit rate (CBR) (percentage of patients who achieve best response of CR, PR or stable disease [SD]).
Duration of response (DoR) | 12 months
  Duration of response (DoR), defined as the time from first documented evidence of CR or PR until disease progression or death.
Time to response (TTR) | 12 months
  Time to response (TTR), defined as the time to the first documented CR or PR.
Progression-free survival (PFS) | 12 months
  Progression-free survival (PFS), defined as the time to disease progression or death due to any cause.
Overall survival (OS) | 12 months
  Overall survival (OS) defined as the time to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Shapira, MD, Principal Investigator — Sheba Medical Center
Locations (6):
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Spain (2):
  - Clínica Universidad de Navarra, Madrid
  - NEXT Madrid, Madrid